CLINICAL TRIAL: NCT01698606
Title: FOR HEALTH: A Family-ORiented Healthy Eating, Activity and Lifestyle Training With Hands-on Experience for Overweight and Obese Preschool Children and Their Families - a Pilot Trial.
Brief Title: FOR HEALTH: A Family-oriented Healthy Eating, Activity and Lifestyle Intervention for Overweight Preschool Children
Acronym: FOR HEALTH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Phase 1 (Feasibility) completed. Currently no funding to launch Phase 2 (RCT).
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Dirk Bock, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 103011
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Childhood Obesity
Keywords: childhood obesity; multidisciplinary; preschool children; community-based; lifestyle intervention; family-centered
MeSH Terms: conditions — Pediatric Obesity | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Secondary lifestyle intervention arm (Active Comparator): 6-month wait list group. Second arm to receive multidisciplinary, family-centered lifestyle intervention with behavioral counseling, following of completion of main 6-month intervention for arm 1.
  Interventions: Behavioral: Multidisciplinary, family-centered lifestyle intervention with behavioral counseling
- Primary lifestyle intervention arm (Experimental): First arm to receive multidisciplinary, family-centered lifestyle intervention with behavioral counseling
  Interventions: Behavioral: Multidisciplinary, family-centered lifestyle intervention with behavioral counseling

INTERVENTIONS:
Behavioral: Multidisciplinary, family-centered lifestyle intervention with behavioral counseling — Parent/caregiver education with skill training and practical activities revolving around healthy dietary choices, establishing an active versus a sedentary lifestyle, and behavioral aspects, while children will be engaged in active play.

SUMMARY:
In this 3-phase study, following an initial small-scale (phase 1) feasibility trial, the aim of phase 2 of the project is to investigate whether a community-based, 12-month intervention for overweight and obese preschool children 2-6 years of age and their families will be effective in reducing the participants' degree of overweight (BMI z-score) and in improving quality of life.

In the final phase (phase 3), participating children will be randomized to either receiving a multidisciplinary lifestyle intervention during the first 6 months (treatment arm), or 6 months later (control or wait list arm), in order to generate more robust effectiveness data. Participants will receive an additional free 6-month YMCA membership while participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-6 on study entry with primary overweight or obesity, BMI => 85th percentile for age and sex on 2010 WHO Growth Charts for Canada
* Family meets Readiness for change criteria, contemplation or higher stage, according to Prochaskas Transtheoretical Model.
* At least one parent/caregiver committed to attend all the program sessions with the child
* Parent/caregiver is agreeing to complete the study questionnaires at the required time points

Exclusion Criteria:

* Chronic medical conditions potentially impacting program participation or associated with a potentially increased risk in participation (e.g. type 1 diabetes mellitus, heart-, gastrointestinal-, or kidney diseases, uncontrolled asthma, other physical, developmental or psychological disabilities that could limit extent of study participation
* Regular use of medications that could limit extent of study participation
* Other concurrent or recently (last 12 months)received obesity treatment
* Inability to read, speak, and/or verbally understand English
* Living outside of the greater London, Ontario, area

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2013-01; Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
BMI z-score | Baseline, 3, 6, 9, 12 months
  Change in BMI z-score

SECONDARY OUTCOMES:
Change in Quality of Life Scores (PedsQL 4.0) | Baseline, 3, 6, 9, 12 months
  Instrument used: PedsQL 4.0 Generic Core Scales, parent report, for toddlers (age 2-4), or for young children (age 5-6).
Change in physical activity score (Netherlands Physical Activity Questionnaire for Young Children, NPAQ) | Baseline, 3, 6, 9, 12 months
Change in parent-reported daily screen-time (TV, computer) | Baseline, 3, 6, 9, 12 months
  Parent-reported daily screen-time, estimated to the nearest 15 minutes.
Change in fruit & vegetable consumption assessed by 3-day food records | Baseline, 3, 6, 9, 12 months
Change in dairy-product consumption assessed by 3-day food records | Baseline, 3, 6, 9, 12 months
Change in grain-product consumption assessed by 3-day food records | Baseline, 3, 6, 9, 12 months
Change in consumption of sugar-sweetened beverages assessed by 3-day food records | Baseline, 3, 6, 9, 12 months
Change in percent overBMI | Baseline, 3, 6, 9, 12 months
  Percent overBMI is the percentage above the 50th percentile of BMI for the respective age and gender [(BMI-BMI at 50th percentile)]/BMI at 50th percentile]*100

OTHER OUTCOMES:
Change in parental BMI (kg/m2) | Baseline, 3, 6, 9, 12 months
  Assessment of change in BMI of the caregiver primary attending the intervention with the child.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk E. Bock, M.D., Principal Investigator — University of Western Ontario, Canada
Locations (1):
- Children's Hospital, London Health Sciences Centre, University of Western Ontario, London, Ontario, Canada